CLINICAL TRIAL: NCT02269748
Title: Patient Morbidity and Root Coverage Outcome After Subepithelial Connective Tissue Graft Used in Combination With Coronally Advanced Flap and Tunneling Technique: a Comparative Randomized Controlled Clinical Trial.
Brief Title: Morbidity and Coverage Outcome With Connective Tissue Graft Used With Coronally Advanced Flap and Tunneling Technique
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Padova, School of Dental Medicine (Other)
Responsible Party: Principal Investigator, Luca Gobbato, Clinical Faculty Department of Periodontology, University of Padova, School of Dental Medicine
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2566P
Record Dates: First submitted 2014-10-15; First posted 2014-10-21 (Estimated); Last update posted 2014-10-21 (Estimated); Status verified 2014-10

CONDITIONS: Gingival Recession
MeSH Terms: conditions — Gingival Recession | interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Root coverage with Tunnel (TT) (Experimental): The tunnel technique with subepithelial connective tissue graft (TT+SeCTG) will be utilized to cover the denude root surface
  Interventions: Procedure: Tunnel technique with subepithelial connective tissue; Drug: Analgesic Therapy
- Coronally advanced flap (CAF+SeCTG) (Active Comparator): The Coronally advanced flap with subepithelial connective tissue graft (CAF+SeCTG) will be utilized to cover the denude root surface
  Interventions: Procedure: Coronally advanced flap; Drug: Analgesic Therapy

INTERVENTIONS:
Procedure: Tunnel technique with subepithelial connective tissue — After harvesting a connective tissue graft from the palate, the graft is placed under a gingival tunnel prepared over the donor site.
  Other Names: root coverage procedure with tunnel technique
  Arms: Root coverage with Tunnel (TT)
Procedure: Coronally advanced flap — After harvesting a connective tissue graft from the palate, the graft is placed under a gingival flap which is repositioned coronally
  Other Names: Coronally advanced flap with sub epithelial connective tissue graft
  Arms: Coronally advanced flap (CAF+SeCTG)
Drug: Analgesic Therapy — Ibuprofen 600 mg TID

SUMMARY:
The aim of this randomized-controlled clinical trial is to compare the patient morbidity and root coverage outcomes of a sub-epithelial connective tissue (SeCTG) used in combination with a coronally advanced flap (CAF) and tunnel technique (TT).

The primary objective of the study is to demonstrate the superiority in terms of the post-operative course and pain of the CAF+SeCTG when compared to the TT.

DETAILED DESCRIPTION:
The aim of this randomized-controlled clinical trial is to compare the patient morbidity and root coverage outcomes of a sub-epithelial connective tissue (SeCTG) used in combination with a coronally advanced flap (CAF) and tunnel technique (TT).

The study will be designed as a single-centre, randomized, clinical trial on the treatment of single gingival recessions. The study assessed two different treatment modalities: the tunnel technique with subepithelial connective tissue graft (TT), compared to the coronally advanced flap with subepithelial connective tissue graft (CAF+SeCTG) in terms of clinical outcomes, and post operative morbidity.

50 patients with one gingival recession each will be treated. Evaluation of patient morbidity will be performed 3 days and 1 week after the surgery. Clinical outcomes will be evaluated 12 months post operatively. Clinical outcomes included percentage of root coverage (RC) and complete root coverage (CRC) will be recorded. Patient morbidity will be evaluated with questionnaires.

Clinical measurements (1 week before surgery and at the 12 months follow-up)

* Gingival recession height (GH)
* Probing depth (PD)
* Clinical attachment level (CAL)
* Height of keratinized tissue (KTH)

Patient morbidity

* Quantity of analgesics taken during the first week post-surgery.
* Patients' post operative discomfort, bleeding, stress and inability to chew was evaluated with a questionnaire given to patients 3 days following surgery.

Kolmogorov-Smirnov test will be used to analyze distribution of continuous variables. Continuous variables are expressed as means ± standard deviation (SD) and compared at baseline by the U Mann-Whitney test. This test will be also used to compare mean changes post vs. baseline measurements. The Wilcoxon test will be used to compare post vs. baseline measurements. Spearman correlation will be used to evaluate associations.

Level of significance was set at 0.05. The SPSS v. 20 software (SPSS Inc., Chicago, IL, USA) will be used for all analyses.

ELIGIBILITY:
Inclusion Criteria:

Single Miller's Class I or Class II recession defects 2 to 4 mm range of recession height will be included presence of identifiable cemento enamel junction (CEJ) presence of a root abrasion, but with an identifiable CEJ, will be accepted; periodontally and systemically healthy no contraindications for periodontal surgery no taking medications known to interfere with periodontal tissue health or healing no periodontal surgery on the involved sites.

Exclusion Criteria:

Subjects smoking more than 10 cigarettes a day will be excluded. Recession defects associated with caries or restoration as well as teeth with evidence of a pulpal pathology will not be included.

Molar teeth will also be excluded.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2012-04; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Patient morbidity | 3 days after intervention
  Quantity of analgesics taken during the first week post-surgery. Patients' post operative discomfort, bleeding, stress and inability to chew was evaluated with a questionnaire given to patients 3 days following surgery.

SECONDARY OUTCOMES:
Clinical measurements GH | 12 months follow-up
  Gingival recession height (GH)
Clinical measurements PD | 12 months follow-up
  Probing depth (PD)
Clinical measurements CAL | 12 months follow-up
  clinical attachment level (CAL)
Clinical measurements KTH | 12 months follow-up
  height of keratinized tissue (KTH)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Padova, Padua, PD, Italy